CLINICAL TRIAL: NCT00066378
Title: An EORTC Randomized, Double Blind, Placebo-Controlled, Phase II Multi-Center Trial Of Anastrozole (Arimidex) In Combination With ZD 1839 (Iressa) Or Placebo In Patients With Advanced Breast Cancer
Brief Title: Anastrozole With or Without Gefitinib in Treating Postmenopausal Women With Metastatic or Locally Recurrent Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EORTC-10021; EORTC-10021; IDBBC-10021
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Gefitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Arimidex + Iressa® 250 mg (Experimental): Arimidex + Iressa® 250 mg Treatment should be administered until documented disease progression, unacceptable toxicity as judged by the responsible physician or patient refusal
  Interventions: Drug: anastrozole; Drug: gefitinib
- Arimidex + Placebo (Active Comparator): Treatment should be administered until documented disease progression, unacceptable toxicity as judged by the responsible physician or patient refusal
  Interventions: Drug: anastrozole

INTERVENTIONS:
Drug: anastrozole
Drug: gefitinib
  Arms: Arimidex + Iressa® 250 mg

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using anastrozole may fight breast cancer by reducing the production of estrogen. Gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Combining anastrozole with gefitinib may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of anastrozole with or without gefitinib in treating postmenopausal women who have metastatic or locally recurrent breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the 1 year antitumor activity of anastrozole with vs without gefitinib, in terms of progression-free survival, in postmenopausal women with metastatic or locally recurrent advanced breast cancer.
* Compare the objective tumor response and duration of tumor response in patients treated with these regimens.
* Compare the progression-free survival of patients treated with these regimens.
* Compare the safety of these regimens in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to participating center, dominant site of metastatic disease (bone alone vs other), prior chemotherapy (no vs yes), stage (metastatic vs locally recurrent), and measurability (measurable vs evaluable). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral anastrozole and oral gefitinib once daily.
* Arm II: Patients receive oral anastrozole and an oral placebo once daily. In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 8 weeks until disease progression.

PROJECTED ACCRUAL: A total of 108 patients (54 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Radiologically or clinically evident metastatic or locally recurrent disease
  * Locally advanced disease in elderly patients
  * Bone metastases only allowed
* Failed prior tamoxifen therapy
* No rapidly progressive visceral metastases
* No uncontrolled CNS metastases
* Hormone receptor status:

  * Estrogen receptor and/or progesterone receptor positive

PATIENT CHARACTERISTICS:

Age

* Postmenopausal

Sex

* Female

Menopausal status

* Postmenopausal, defined by any of the following:

  * Natural menopause with last menses more than 1 year ago
  * Radiotherapy-induced oophorectomy with last menses more than 1 year ago
  * Chemotherapy-induced menopause with last menses more than 1 year ago AND serum follicle-stimulating hormone and luteinizing hormone and plasma estradiol levels clearly in the postmenopausal range
  * Surgical castration

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Transaminases no greater than 2.5 times ULN
* No unstable or uncompensated hepatic disease

Renal

* No unstable or uncompensated renal disease

Cardiovascular

* No unstable or uncompensated cardiac disease

Pulmonary

* No unstable or uncompensated pulmonary disease
* No clinically active interstitial lung disease

  * Asymptomatic chronic stable radiographic changes are allowed

Other

* No severe or uncontrolled systemic disease
* No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix, nonmelanoma skin cancer, or contralateral breast cancer
* No psychological, familial, sociological or geographical condition that would preclude study compliance and follow-up
* No grade 2 or greater unresolved chronic toxicity from prior anticancer therapy
* No unresolved ocular inflammation or infection
* No known hypersensitivity to anastrozole or gefitinib or any of their excipients

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior trastuzumab (Herceptin)
* No concurrent biologic therapy

Chemotherapy

* No more than 1 line of prior chemotherapy in the adjuvant or metastatic setting
* No concurrent chemotherapy

Endocrine therapy

* At least 2 years since prior aromatase inhibitors (e.g., anastrozole, letrozole, or exemestane) in the adjuvant setting
* Prior tamoxifen or fulvestrant in the adjuvant and/or metastatic setting allowed
* No prior aromatase inhibitors for metastatic disease
* No other concurrent hormonal therapy

Radiotherapy

* No concurrent radiotherapy to any metastatic site

Surgery

* No surgery during and within 4 days after the last dose of gefitinib

Other

* At least 30 days since prior investigational drugs
* No prior anti-epidermal growth factor therapy
* No prior anti-vascular endothelial growth factor therapy (i.e., tyrosine kinase inhibitor receptor)
* No concurrent administration of any of the following drugs:

  * Phenytoin
  * Carbamazepine
  * Rifampin
  * Phenobarbital
  * Hypericum perforatum (St John's Wort)
* No other concurrent investigational drugs or treatment
* No other concurrent cancer treatment
* No concurrent systemic retinoids
* Concurrent bisphosphonate therapy for the treatment and prevention of bony metastases is allowed provided therapy was initiated prior to study entry

  * Bisphosphonates may be initiated during study only for the treatment of hypercalcemia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2003-05; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 1 year | at 1 year

SECONDARY OUTCOMES:
Tumor response as measured by RECIST | from randomisation
Duration of response as measured by RECIST | response duration
Safety as measured by CTC v2.0 | from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Martine J. Piccart, MD, PhD, Study Chair — Jules Bordet Institute
Locations (9):
- Belgium (3):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Algemeen Ziekenhuis Sint-Augustinus, Wilrijk
- France (2):
  - Institut Bergonie, Bordeaux
  - Centre Henri Becquerel, Rouen
- Netherlands (2):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
- Institute of Oncology - Ljubljana, Ljubljana, Slovenia
- Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Result] Mauriac L, Cameron D, Dirix L: Results of randomized phase II trial combining Iressa (gefitinib) and arimidex in women with advanced breast cancer (ABC): EORTC protocol 10021. [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-6133, 2008.
- [Derived] Tryfonidis K, Basaran G, Bogaerts J, Debled M, Dirix L, Thery JC, Tjan-Heijnen VC, Van den Weyngaert D, Cufer T, Piccart M, Cameron D; EORTC-Breast Cancer Group. A European Organisation for Research and Treatment of Cancer randomized, double-blind, placebo-controlled, multicentre phase II trial of anastrozole in combination with gefitinib or placebo in hormone receptor-positive advanced breast cancer (NCT00066378). Eur J Cancer. 2016 Jan;53:144-54. doi: 10.1016/j.ejca.2015.10.012. Epub 2015 Dec 24. PMID 26724641